CLINICAL TRIAL: NCT02973451
Title: Laparoscopic Guided Transversus Abdominis Plane Block Versus Trocar Site Local Anesthetic Infiltration in Gynecologic Laparoscopy.
Brief Title: Laparoscopic Guided Transversus Abdominis Plane Block Versus Trocar Site Infiltration in Gynecologic Laparoscopy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2016-11

CONDITIONS: Post Operative Local Anaesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic (Active Comparator): Laparoscopic Guided Transversus Abdominis Plane Block using Bupivacaine
  Interventions: Drug: Laparoscopic Guided Bupivacaine
- local (Active Comparator): Trocar Site Infiltration of Bupivacaine
  Interventions: Drug: local Bupivacaine

INTERVENTIONS:
Drug: Laparoscopic Guided Bupivacaine — Bupivacaine Laparoscopic GuidedTransversus Abdominis Plane Block
  Other Names: marcaine
  Arms: Laparoscopic
Drug: local Bupivacaine — Bupivacaine Trocar Site Infiltration
  Other Names: marcaine
  Arms: local

SUMMARY:
to compare between Laparoscopic Guided Transversus Abdominis Plane Block and Trocar Site Infiltration as postoperative analgesia in Gynecologic Laparoscopic surgery.

DETAILED DESCRIPTION:
two groups of patients who are eligible for Gynecologic Laparoscopy were randomized to either Laparoscopic Guided Transversus Abdominis Plane Block or Trocar Site Infiltration at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* patients Need Gynecologic Laparoscopy

Exclusion Criteria:

* diagnosed with chronic pain syndrome
* have a postoperative intraperitoneal drain
* necessitating alteration to laparotomy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A el sharkwy, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt